CLINICAL TRIAL: NCT02598726
Title: Phase 1 Pilot Study of Curcumin and Piperine to Derive a Safe, Optimal Biologic Dose for Ureteral Stent-Induced Symptoms in Cancer Patients
Brief Title: Curcumin and Piperine in Reducing Inflammation for Ureteral Stent-Induced Symptoms in Patients With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC1511; NCI-2015-01716 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1511 (Other: Mayo Clinic); UG1CA189823 (NIH); 15-003188 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2015-10-14; First posted 2015-11-06 (Estimated); Last update posted 2025-04-22 (Actual); Status verified 2024-11

CONDITIONS: Bladder Spasm; Malignant Neoplasm; Pain; Urinary Urgency
MeSH Terms: conditions — Neoplasms; Pain | interventions — Curcumin; piperine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (curcumin, piperine) (Experimental): Patients receive curcumin PO BID or TID and piperine extract (standardized) PO on days 1-7 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Curcumin; Other: Laboratory Biomarker Analysis; Dietary Supplement: Piperine Extract (Standardized); Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Curcumin — Given PO
  Other Names: C.I. 75300; C.I. Natural Yellow 3; Diferuloylmethane; Turmeric Yellow
Other: Laboratory Biomarker Analysis — Correlative studies
Dietary Supplement: Piperine Extract (Standardized) — Given PO
  Other Names: Bioperine; Standardized Piperine Extract
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase I trial studies the side effects and best dose of curcumin when given together with piperine (piperine extract [standardized]) in reducing inflammation for ureteral stent-induced symptoms in patients with cancer. Curcumin is a spice similar to turmeric and works by decreasing the chemical moderators that produce inflammation in the body. Piperine is pepper and works by increasing the amount of curcumin available in the body when taken with curcumin. Giving curcumin together with piperine may reduce inflammation and discomfort from a ureteric stent in older patients with cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a dose-escalation study with curcumin and piperine to derive a safe, optimal biological dose of this combination in cancer patients.

SECONDARY OBJECTIVES:

I. To describe the grade 2+ toxicities associated with curcumin and piperine. II. To evaluate quality of life associated with this combination by means of the Mayo Modified Urinary Stent Symptom Questionnaire (USSQ).

TERTIARY OBJECTIVES:

I. To characterize the change in urinary prostaglandin E2 concentrations that occur at baseline and then after one week of curcumin + piperine.

OUTLINE: This is a dose-escalation study of curcumin.

Patients receive curcumin orally (PO) twice daily (BID) or thrice daily (TID) and piperine extract (standardized) PO on days 1-7 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Ureteral stent in place at study registration
* Patient reports pain, spasms, or urgency symptoms after stent placement, which are thought to be unrelated to other causes as per the patient or healthcare provider or both (documentation in the medical record is unnecessary)
* Ability to complete English language questionnaires by themselves or with assistance
* After the week-long study treatment, participants must be willing to return to the enrolling institution for a follow-up visit
* Willingness to provide mandatory 24 hour urine collection samples for research purposes
* Able to swallow supplements
* Patient must have either a history of cancer or active cancer
* Registration >= 7 days after placement of a new stent or >= 3 days after a stent exchange
* Willingness to refrain from grapefruit juice for 7 days prior to and for 7 days during the study

Exclusion Criteria:

* Receiving warfarin at registration
* Active cholecystitis
* Taking any of the following drugs at the time of study participation: epidermal growth factor receptor inhibitor, topoisomerase 1 inhibitor (camptothecin, irinotecan); buspirone, benzodiazepines, zolpidem, calcium channel blockers (such as felodipine, nifedipine, verapamil); digoxin or quinidine; codeine or fentanyl; phenytoin, propranolol, rifampin, or theophylline
* History of alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, using the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 1 month post-treatment
  Examined in an exploratory and hypothesis-generating fashion. The number and severity of all adverse events (overall, by dose-level, and by tumor type) will be tabulated and summarized in this patient population. The grade 2+ adverse events will also be described and summarized in a similar fashion.
Maximum tolerated dose (MTD) of curcumin in combination with piperine | 7 days
  The MTD of curcumin in combination with piperine is defined as the highest safely tolerated dose level where at most 1 out of 6 patients experience a dose limiting toxicity (DLT) with the next higher dose having at least 2 patients out of a maximum of 6 patients experiencing a DLT. DLT will be assessed using Common Terminology Criteria for Adverse Events version 4.0. Examined in an exploratory and hypothesis-generating fashion.
Optimal biologically active dose for curcumin in combination with piperine extract (standardized) | 7 days
  Examined in an exploratory and hypothesis-generating fashion.

SECONDARY OUTCOMES:
Change in quality of life (QOL) by means of the USSQ | Baseline to 7 days
  Reported descriptively. Graphical methods and descriptive statistics will be used to describe the QOL data at baseline and after treatment. Change in QOL from baseline will be assessed via the paired t-test or non-parametric equivalent (Wilcoxon Signed-Rank test). The questions from the USSQ will be summarized descriptively via frequency tables.

OTHER OUTCOMES:
Change in prostaglandin E2 concentrations | Baseline to 7 days
  Graphical methods and descriptive statistics will be used to summarize the prostaglandin E2 concentration data. This will be done overall and by dose level. Changes will be summarized by reporting the mean and median percent change from baseline to post-treatment. Percent and absolute change from baseline will also be assessed using the Wilcoxon Signed-Rank test. Fisher's Exact test will be used for assessing the association between categorical variables and the t-test will be used for comparing prostaglandin E2 concentration data across different patient subgroups of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials